## STATISTICAL ANALYSIS PLAN

Study Title: Determining the Effect of Music on Pain, Anxiety and Vital Signs in Cancer

Patients Treated in Palliative Care Centers: A Quasi-Experimental Study

**Unique Protocol ID: KMU-SHMYO-GK-01** 

NCT Number: .....

**Document Date: November 1, 2022** 

Principal Investigator: Gülsüm Kehribar, PhD

Institution: Karamanoğlu Mehmetbey University

**Ethics Committee Approval Number: 2021.01/06** 

**Ethics Committee Approval Date: 27.01. 2021** 

Ethics Committee: Yozgat Bozok University Invasive (Non-Interventional) Clinical

**Research Ethics Committee** 

Evaluation of Data: Statistical analyses were performed using SPSS version 24 (Statistical Package For Social Sciences) software. The conformity of the variables to the normal distribution was examined using visual (histogram and probability graphs) and analytical methods (Shapiro-Wilk Test). Descriptive analyses are given using the mean and standard deviation for normally distributed variables. Number and % are given for nominal variables. The T-test was used in independent groups to compare the measured values of the intervention and control groups.

The Chi-Square Test (Pearson Chi-Square) was used to compare the intervention and control groups for categorical variables. Two-Way Analysis of Variance (Mixed Design-Repeated Measurement ANOVA) was used in repeated measurements to evaluate the change over time of the measured variables of the intervention and control groups and their group-time interactions. The statistical significance level was accepted as p<0.05.